CLINICAL TRIAL: NCT05179317
Title: A Phase II Study of QL1706 Plus Chemotherapy With or Without Bevacizumab for the First-Line Treatment of Recurrent, or Metastatic Cervical Cancer
Brief Title: Safety and Efficacy Study of First-line Treatment With QL1706 Plus Chemotherapy With or Without Bevacizumab in Women With Recurrent, or Metastatic Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-204
Record Dates: First submitted 2021-12-09; First posted 2022-01-05 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2021-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706+chemotherapy±Bevacizumab (Experimental): On Day 1 of each 21-day cycle, participants receive an intravenous (IV) infusion of QL1706 5mg/kg plus Investigator choice of chemotherapy (paclitaxel 175 mg/m^2 plus cisplatin 70 mg/m^2 or paclitaxel 175 mg/m^2 plus carboplatin Area Under the Curve (AUC) 6 withor without bevacizumab 15 mg/kg)
  Interventions: Drug: QL1706

INTERVENTIONS:
Drug: QL1706 — Drug: QL1706 Intravenous Infusion
  Drug: Paclitaxel injection Intravenous Infusion
  Drug: Cisplatin/Carboplatin Intravenous Infusion
  Drug:Bevacizumab Intravenous Infusion

SUMMARY:
This is a Phase 2, multicenter, open label, single arm study designed to evaluate the efficacy, safety, tolerability, pharmacokinetic (PK), and immunogenicity of QL1706 Plus Chemotherapy in Women With Recurrent, or Metastatic Cervical Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of study entry.
2. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Life expectancy of at least 12 weeks.
4. At least one measurable lesion (according to RECIST v1.1)
5. Cervical squamous cell carcinoma, adenocarcinoma and adenosquamous cell carcinoma diagnosed by histopathology and confirmed by imaging as recurrent or stage ⅣB cervical cancer.
6. No brain metastasis, or no meningeal metastasis.
7. Patients must have normal function as defined:
8. Any unresolved AEs ≤ CTCAE Grade 1 (except alopecia).
9. Negative pregnancy test for females of child-bearing potentials.
10. Patients with reproductive function agreed to take effective contraceptive measures during the treatment and in 6 months after the end of administration.
11. Patients must be able to understand and volunteer to sign the informed consent.

Exclusion Criteria:

1. Has received prior chemoradiotherapy within 3 months before enrollment,or has received prior radiotherapy within 2 weaks before enrollment.
2. Is currently participating in or has participated in a study of an investigational agent within 4 weeks before enrollment.
3. Has any active autoimmune diseases or a history of autoimmune diseases (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid hyperfunction; patients with vitiligo; complete remission of asthma in childhood, can be included without any intervention after adulthood; asthma patients who require bronchodilators for medical intervention cannot be included).
4. Is using immunosuppressive agents or systemic hormonal therapy to achieve immunosuppressive purposes (agents amount > 10 mg / day of prednisone or other therapeutic hormones), and continue to use within 2 weeks before enrollment.
5. Known history of hypersensitivity to macromolecular protein preparation or any components of the QL1604 formulation, or any components of the study drugs.
6. Has uncontrolled clinically significant cardiac and cerebral vascular diseases within 6 months before enrollment, including but not limited to the following: myocardial infarction, severe or unstable angina, coronary artery/peripheral artery bypass grafting, congestive heart failure, cerebrovascular accident (including transient ischemic attack).
7. Symptomatic congestive heart failure (New York Heart Association Grade II-IV), or NCI-CTCAE v5.0 ≥ 2 arrhythmia, atrial fibrillation of any grade, or clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention.
8. Has active infection or an unexplained fever > 38.5°C during screening visits( subjects with tumor fever may be enrolled at the discretion of the investigator).
9. Hepatitis b surface antigen (HBsAg) positive and/or hepatitis b core antibody (HBcAb) positive and HBVDNA>103copies/ml, hepatitis c virus antibody positive .
10. Known history of human immunodeficiency virus (HIV) infection, or other acquired or congenital immunodeficiency diseases,or has a history of organ transplantation (except corneal transplantation).
11. Has been vaccinated with live anti-tumor vaccine, or have received anti-tumor immunotherapy, or may receive other systemic anti-tumor treatments during the study period.
12. Has a clear history of neurological or mental disorders, including epilepsy or dementia.
13. Patients with other malignancies witnin 5 years( except cured basal cell carcinoma of skin cancer, papillary thyroid carcinoma).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced At Least One Adverse Event (AE) | Up to approximately 2 years
  An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of all participants who experienced at least one AE is presented.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shangdong

REFERENCES:
- [Derived] Zhao Y, Ma Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Hao Y, Chen J, Zhang G, Qu S, Li Y, Feng W, Yang M, Liu B, Ouyang W, Liang J, Yu Z, Kang X, Xue S, Yang G, Yan W, Yang Y, Liu Z, Peng Y, Fanslow B, Huang X, Zhang L, Zhao H. First-in-human phase I/Ib study of QL1706 (PSB205), a bifunctional PD1/CTLA4 dual blocker, in patients with advanced solid tumors. J Hematol Oncol. 2023 May 8;16(1):50. doi: 10.1186/s13045-023-01445-1. PMID 37158938